CLINICAL TRIAL: NCT02085343
Title: Anti-phobic and Safety Behaviors in the Treatment of Acrophobia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2013-02-0023
Record Dates: First submitted 2014-01-22; First posted 2014-03-12 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Specific Phobia
Keywords: Exposure therapy; Specific phobia; Fear of heights; Acrophobia; Safety behavior fading; Anti-phobic Actions
MeSH Terms: conditions — Phobia, Specific; Acrophobia | interventions — Implosive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- EXP + SBF + AA (Experimental): Exposure therapy (EXP) with safety behavior fading (SBF) and anti-phobic action (AA)
  Interventions: Behavioral: EXP; Behavioral: EXP + SBF; Behavioral: EXP + SBF + AA
- EXP + SBF (Active Comparator): Exposure therapy (EXP) with safety behavior fading (SBF)
  Interventions: Behavioral: EXP; Behavioral: EXP + SBF
- EXP (Active Comparator): Standard therapist-guided in vivo exposure therapy (EXP)
  Interventions: Behavioral: EXP
- Wait-list control (No Intervention): Subjects assigned to this arm will undergo assessments at Weeks 0, Week 1, and Week 5, but will not receive any interventions.

INTERVENTIONS:
Behavioral: EXP — Participants will receive one-session exposure therapy consisting of six-6 minute trials of exposure to heights, involving ascending a 9-landing flight of outdoor stairs. Participants will be asked to ascend, accompanied by the therapist who will provide verbal encouragement throughout supporting efforts at exposure. An instructional set will be provided prior to treatment presenting the rationale for exposure as an effective means of reducing pathological fear.
  Other Names: Standard Therapist-Guided In Vivo Exposure Therapy (EXP)
  Arms: EXP; EXP + SBF; EXP + SBF + AA
Behavioral: EXP + SBF — Participants will receive one-session exposure therapy consisting of six-6 minute trials of exposure to heights, involving ascending a 9-landing flight of outdoor stairs. Participants will be asked to ascend, accompanied by the therapist who will provide verbal encouragement supporting efforts at exposure. An instructional set will be provided prior to treatment explaining how safety behaviors serve to maintain fear, and how their elimination may enhance fear reduction. Additionally, the therapist will identify safety behaviors and prompt participants to reduce their utilization of them during treatment.
  Other Names: Exposure Therapy with Safety Behavior Fading (EXP + SBF)
  Arms: EXP + SBF; EXP + SBF + AA
Behavioral: EXP + SBF + AA — Participants will receive one-session exposure therapy consisting of six-6 minute trials of exposure to heights, involving ascending a 9-landing flight of outdoor stairs. Participants will be asked to ascend, accompanied by the therapist who will provide verbal encouragement supporting efforts at exposure. An instructional set will be provided explaining the rationale for eliminating safety behaviors, and how engagement in anti-phobic actions may enhance fear reduction. Additionally, the therapist will identify safety behaviors and prompt participants to reduce their utilization of them during treatment, and will instruct participants to enact a series of progressively challenging anti-phobic actions which oppose the prototypical fear response.
  Other Names: Exposure with Safety Behavior Fading and Anti-Phobic Actions
  Arms: EXP + SBF + AA

SUMMARY:
This study tests whether a single session of exposure therapy may be enhanced by the addition of anti-phobic actions beyond the mere fading of safety behaviors. A total of 100 acrophobic participants will be randomly assigned to receive standard exposure therapy (EXP), exposure therapy with safety behavior fading (EXP + SBF), exposure with safety behavior fading and anti-phobic actions (EXP + SBF + AA), or to a wait-list control group (WL).

DETAILED DESCRIPTION:
This study tests whether a single session of exposure therapy may be enhanced by the addition of one of two augmentation strategies, including engagement in anti-phobic actions and fading of safety behaviors. Because utilization of safety behaviors is functionally precluded by anti-phobic action, the present study design will both replicate and extend prior research by addressing whether anti-phobic actions enhance exposure therapy beyond the mere fading of safety behaviors. A total of 100 individuals between the ages of 18 and 65 meeting DSM-IV criteria for acrophobia (fear of heights) will be randomly assigned to one of four conditions including (1) standard exposure therapy, (2) exposure therapy with safety behavior fading, (3) exposure therapy with safety behavior fading and anti-phobic actions, and (4) a wait-list control condition. All participants will complete an online prescreen and face-to-face screening assessment to determine eligibility and pre-treatment symptom severity. Participants will also complete assessments at post-treatment and 1-month follow-up assessments. Subjective fear during two behavioral approach tests (in the treatment and generalization context, respectively) conducted at pre-treatment, post-treatment, and 1-month follow-up assessments will serve as the primary measure of treatment outcome. Additionally, a battery of self-report questionnaires will be completed at pre-treatment, during treatment, at post-treatment, and at a 1-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65.
2. Fluent in English (written and spoken). This is required because assessment instruments are validated only in English.
3. Meet DSM-IV criteria for specific phobia, natural environment type, with acrophobic concerns, based on the Composite International Diagnostic Interview (CIDI-Auto; World Health Organization, 1997).
4. Report moderate fear or avoidance (i.e., a score of 30 or higher) on a modified version of the Acrophobia Questionnaire (AQ; Cohen, 1977).
5. Exhibit at least moderate fear (i.e., a fear score of 50 or higher, where 0 = no fear and 100 = extreme fear) during two behavioral approach tests (BATs) consisting of ascending two moderately challenging flights of stairs.

Exclusion Criteria:

1. Medical condition(s) which may prevent safely climbing or descending stairs or walking for more than 15 minutes at a time (It will be necessary to walk to different sites for the behavioral approach tests).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-02; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Peak subjective fear (0 - 100) upon exposure to heights in the generalization context. | Pre-treatment (1 week before treatment), treatment (1 week after pre-treatment), post-treatment (immediately following treatment), and follow-up (1 month after treatment).
  Peak subjective fear ratings (0 - 100).

SECONDARY OUTCOMES:
Acrophobia Questionnaire - Modified (Cohen, 1977; Wolitzky & Telch, 2009) | Pre-treatment (1 week before treatment), treatment (1 week after pre-treatment), post-treatment (immediately following treatment), and follow-up (1 month after treatment).
  20-item Likert-type scale assessing acrophobic symptoms
Height estimation task | Pre-treatment (1 week before treatment), treatment (1 week after pre-treatment), post-treatment (immediately following treatment), and follow-up (1 month after treatment).
  Perceptual task requiring estimation of height from the top of a flight of stairs
Heart rate | Pre-treatment (1 week before treatment), treatment (1 week after pre-treatment), post-treatment (immediately following treatment), and follow-up (1 month after treatment).
  Heart rate reactivity assessed using a Polar Heart Rate Monitor.
Treatment Process Questionnaire | Treatment (1 week following pre-treatment assessment)
  Self-efficacy, anticipated anxiety, anticipated danger, and utilization of safety behaviors assessed via self-report.

CONTACTS AND LOCATIONS:
Overall Officials: Adam R. Cobb, MA, Study Director — The University of Texas at Austin; Michael J. Telch, PhD, Principal Investigator — The University of Texas at Austin
Locations (1):
- The University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be shared upon request to the corresponding investigator / author upon project completion. Contact Michael J. Telch, Ph.D at telch@austin.utexas.edu